CLINICAL TRIAL: NCT04318938
Title: Advancing Brigatinib Properties in Anaplastic Lymphoma Kinase Positive Non-small Cell Lung Cancer (ALK+ NSCLC) Patients
Brief Title: Advancing Brigatinib Properties in ALK+ NSCLC Patients by Deep Phenotyping
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Thoraxklinik-Heidelberg gGmbH (Other); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABP
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: NSCLC
Keywords: ALK+ NSCLC; Resistance patterns; Molecular properties
MeSH Terms: interventions — brigatinib; Pharmaceutical Preparations; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm with any available ALK TKI (Active Comparator): 1. st line: Any approved 2nd-generation TKI according to investigator's choice
  2. nd line: Any available ALK TKI according to investigator's choice (patients from the standard Arm A can be offered brigatinib in the 2nd line)
  Interventions: Drug: Tyrosine kinase inhibitor
- Experimental Arm with Brigatinib (Experimental): 1. st line: 90 mg brigatinib once daily p.o. for the first 7 days (lead-in) followed by 180 mg brigatinib once daily p.o. afterwards, starting with day 8
  2. nd line: Any available ALK TKI according to investigator's choice
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Treatment with Brigatinib
  Other Names: Study treatment
  Arms: Experimental Arm with Brigatinib
Drug: Tyrosine kinase inhibitor — Treatment with any TKI
  Other Names: Study treatment
  Arms: Standard Arm with any available ALK TKI

SUMMARY:
This is a prospective, randomized, open-label, multicenter phase II study investigating the advancing Brigatinib properties in anaplastic lymphoma kinase positive non-small cell lung cancer (ALK+ NSCLC) patients by deep phenotyping

DETAILED DESCRIPTION:
The aim of this study is to compare efficacy of brigatinib and other 2nd-generation ALK tyrosin kinase inhibitor (TKI) in 1st and 2nd line treatment and to explore resistance patterns according to treatment and molecular properties of the tumors

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed written consent and any locally-required authorization (EU Data Privacy Directive) given by the patient
2. Male or female ≥ 18 years of age NOTE: There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
3. Histologically confirmed locally advanced (stage III) and not suitable for curative treatment, i.e. R0 operation or definitive chemo-/radiation, or metastatic (stage IV) ALK+ NSCLC NOTE: Documentation of ALK rearrangement by a positive result of any ALK assay approved in Germany [i.e. positivity for at least one of the three: immunohistochemistry (IHC), NGS, fluorescence in situ hybridisation (FISH)] must be available at baseline. Treatment can already be started based on a local ALK+ test result, but subsequent central testing of the baseline biopsy for molecular profiling, incl. determination of ALK variant and TP53 status, should be made possible for all patients.
4. No prior therapy for metastatic ALK+ NSCLC including therapy with ALK inhibitors. However, 1 or 2 cycles of chemotherapy, chemo-immunotherapy or immunotherapy as well as cerebral irradiation before inclusion in the study will be allowed.
5. At least 1 measurable (i.e., target) lesion per RECIST v1.1 or otherwise evaluable lesion (e.g. brain lesion with at least 5 mm of longest diameter if measured by high-resolution cMRT e.g. using 1 mm slices thickness and not planned for irradiation before the first response assessment).
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
7. Have adequate organ function, as determined by:

   * Total bilirubin ≤1.5x the upper limit of the normal range (ULN) (< 3x the ULN if Gilbert's disease is present)
   * Estimated glomerular filtration rate ≥30 mL/minute/1.73 m2 (calculated by Modification of Diet in Renal Disease (MDRD) or any other validated formula, see Appendix 13.4)
   * Alanine aminotransferase/aspartate aminotransferase ≤2.5x ULN NOTE: ≤5x ULN is acceptable if liver metastases are present.
   * Serum lipase or serum amylase ≤ 1.5x ULN
   * Platelet count ≥75x 109/L
   * Hemoglobin ≥9 g/dL
   * Absolute neutrophil count ≥1.5x 109/L
8. Willingness and ability to comply with scheduled visit and study procedures
9. Patient willing to participate in accompanying research program
10. Collection of current biopsy during screening must be feasible NOTE: For each patient a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block must be available for biomarker evaluation. Excisional, incisional or core needle biopsies are appropriate, while fine needle aspirations are insufficient.
11. Women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days prior to randomization. Women must not be breastfeeding.
12. Female patients who:

    * are postmenopausal for at least 1 year before the screening visit, OR
    * are surgically sterile, OR
    * if they are of childbearing potential, agree to practice highly effective non-hormonal contraception from the time of signing the informed consent through at least 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.

Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

* agree to practice effective barrier contraception during the entire study treatment period and through at least 3 months after the last dose of study drug, OR
* agree to completely abstain from heterosexual intercourse.

Exclusion Criteria:

1. History or presence at baseline of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis
2. Uncontrolled hypertension, defined as hypertension treated* with anti-hypertensive drugs AND blood pressure ≥ 160 mmHg (systolic) or ≥ 100 mmHg (diastolic) in repeated measurements. Untreated elevated blood pressure is not an exclusion criterion and should receive adequate anti-hypertensive adjustment.

   *Please notecase of treatment, at least 3 anti-hypertensive drugs should have been used with the intention to control hypertensive disease
3. Systemic treatment with strong cytochrome P-450 (CYP) 3A inhibitors, strong CYP3A inducers, or moderate CYP3A inducers or treatment with any investigational systemic anticancer agents, chemotherapy or radiation therapy (except for stereotactic radiosurgery or stereotactic radiation therapy or palliative radiotherapy) within 14 days of randomization
4. Treatment with antineoplastic monoclonal antibodies within 30 days of randomization
5. Major surgery within 30 days of randomization. Minor surgical procedures, such as catheter placement or minimally invasive biopsies, are allowed.
6. Current symptomatic spinal cord compression as confirmed by radiographic imaging. Patients with leptomeningeal disease without symptomatic cord compression are allowed.
7. Significant or uncontrolled cardiovascular disease, defined as to the following:

   * If an acute myocardial infarction has ensued in the past 6 months, successful reperfusion has to be documented and the patient has to be free of symptoms
   * New York Heart Association Class III or IV heart failure (i.e. marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest) within 6 months prior to randomization
   * Any history of clinically significant ventricular arrhythmia, defined as ventricular tachycardia (VT), ventricular fibrillation (VF), or cardiac arrest
8. Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose of study drug
9. Malabsorption syndrome or other gastrointestinal illness or condition that could affect oral absorption of the study drug
10. Active severe or uncontrolled chronic infection, including but not limited to, the requirement for intravenous antibiotics for longer than 2 weeks
11. History of HIV infection. Testing is not required in the absence of history.
12. Chronic hepatitis B (surface antigen-positive) or chronic active hepatitis C infection. Testing is not required in the absence of history.
13. Any serious medical condition or psychiatric illness that could, in the investigator's opinion, potentially compromise patient safety or interfere with the completion of treatment according to this protocol
14. Known or suspected hypersensitivity to brigatinib or other TKI or their excipients
15. Life-threatening illness unrelated to cancer
16. Involvement in the planning and/or conduct of the study (applies to both Takeda staff and/or staff of sponsor and study site)
17. Patient who might be dependent on the sponsor, site or the investigator
18. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities [according to national Medicinal Products Act (Arzneimittelgesetz, AMG)]
19. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [according to national AMG]
20. Legal incapacity or limited legal capacity
21. Females who are pregnant or breastfeeding
22. Patients who have symptomatic CNS metastases (parenchymal or leptomeningeal) at screening or asymptomatic disease requiring an increasing dose of corticosteroids to control symptoms within 7 days prior to randomization.

    NOTE: If a patient has worsening neurological symptoms or signs due to CNS metastasis, the patient needs to complete local therapy and be neurologically stable (with no requirement for an increasing dose of corticosteroids or use of anticonvulsants) for 7 days prior to randomization.
23. Rare hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of 1st-line treatment according to RECIST v1.1 | 68 months
  Time from the first dosing date of any study medication to the date of the first objectively documented tumor progression or death due to any cause

SECONDARY OUTCOMES:
PFS of 2nd-line treatment according to RECIST v1.1 | 68 months
  Time from the first dosing date of any 2nd-line TKI to the date of the objectively documented tumor progression or death due to any cause
TNT 1st line (TNT1, i.e. time-to-next treatment for the 1st line) | 68 months
  Time from begin of 1st-line treatment until begin of 2nd-line treatment
TNT 2nd line (TNT2, i.e. time-to-next treatment for the 2nd line | 68 months
  Time from begin of 2nd line until begin of 3rd-line treatment
TNT1/2 (time-to-next treatment for the 1st and 2nd line together) | 68 months
  Time from begin of 1st-line treatment until begin of 3rd-line treatment
Overall survival (OS) | 68 months
  Time from treatment start in the 1st line to the date of death (due to any cause)
Intracranial ORR (iORR) | 68 months
  Percentage of participants with a best overall intracranial response (BOR) of intracranial complete response (CR) or intracranial partial response (PR). Best overall intracranial response (BOR) is defined as the best response designation, recorded between the date of first dose and the date of the initial objectively documented intracranial tumor progression per RECIST criteria or the date of subsequent therapy or death, whichever occurs first.
Intracranial DOR (iDOR) according to RECIST v1.1 | 68 months
  Time from first documentation of intracranial CR or PR according to RECIST v1.1 (whichever is first recorded) until the first date that the intracranial progressive disease (PD) is objectively documented or until death (whichever occurs first
Time to intracranial progression (TTiP) | 68 months
  Time from start of 1st-line treatment until the occurrence of a new central nervous system (CNS) lesion or progression of pre-existing CNS lesions
Safety (rate of adverse events) | 68 months
  Type, incidence and severity of adverse events (AEs) and serious adverse events (SAEs)graded according to NCI CTCAE v5.0
Quality of life (QoL) assessed by SF-12-questionnaire | 68 months
  Patient reported outcome assessed by the validated SF-12-questionnaire
Quality of life (QoL) assessed by EORTC-quality of life questionnaire (QLQ)-BN20-questionnaire | 68 months
  Patient reported outcome assessed by the validated EORTC-QLQ-BN20-questionnaire

OTHER OUTCOMES:
ALK variant analysis in tumor tissue | 68 months
  Typing of ALK fusion variants in tumor samples
ALK variant analysis in blood samples | 68 months
  Typing of ALK fusion variants in blood samples
TP53 mutation status in tumor tissue | 68 months
  Assessment of TP53 mutation status in tumor samples
TP53 mutation status in blood samples | 68 months
  Assessment of TP53 mutation status in blood samples
Detection of "acquired resistance" mutations in tumor tissue | 68 months
  Detection of "acquired resistance" mutations via standardized next-generation sequencing (NGS)-based multiplex analysis in tumor samples
Detection of "acquired resistance" mutations in blood samples | 68 months
  Detection of "acquired resistance" mutations via standardized next-generation sequencing (NGS)-based multiplex analysis in blood samples
ALK variant analysis in cerebrospinal fluid | 68 months
  Typing of ALK fusion variants in cerebrospinal fluid in "brain-only" progression.
TP53 mutation status in cerebrospinal fluid | 68 months
  Assessment of TP53 mutation status in cerebrospinal fluid in "brain-only" progression.
Detection of "acquired resistance" mutations in cerebrospinal fluid | 68 months
  Detection of "acquired resistance" mutations via standardized circulating tumor DNA (ctDNA) next-generation sequencing (NGS)-based multiplex analysis in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Study Director — Institut für Klinische Krebsforschung IKF GmbH
Locations (26):
- Germany (26):
  - HELIOS Klinikum Emil von Behring, Berlin
  - Charité Berlin, Berlin
  - Lungenklinik Köln - Merheim, Cologne
  - Universitätsmedizin Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Niels-Stensen-Kliniken Georgsmarienhütte, Georgsmarienhütte
  - Universitätsklinikum Gießen, Giessen
  - Studiengesellschaft Hämato-Onkologie Hamburg, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - KRH Klinikum Siloah Hannover, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Klinik der LMU München - Innenstadt, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Pius Hospital Oldenburg, Oldenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Klinik Schillerhöhe, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Christopoulos P, Bozorgmehr F, Bruckner L, Chung I, Krisam J, Schneider MA, Stenzinger A, Eickhoff R, Mueller DW, Thomas M. Brigatinib versus other second-generation ALK inhibitors as initial treatment of anaplastic lymphoma kinase positive non-small cell lung cancer with deep phenotyping: study protocol of the ABP trial. BMC Cancer. 2021 Jun 28;21(1):743. doi: 10.1186/s12885-021-08460-w. PMID 34182952